CLINICAL TRIAL: NCT02713295
Title: A Non-interventional Prospective Cohort Study to Provide Real-world Evidence on the Treatment Goal Achievement Rate, Adherence to and Utilization Patterns of Adalimumab in Patients With Moderate to Severe Plaque Psoriasis in Greece
Brief Title: A Study to Provide Real-world Evidence on the Treatment Goal Achievement Rate, Adherence to and Utilization Patterns of Adalimumab in Patients With Moderate to Severe Plaque Psoriasis in Greece
Acronym: CONCORDIA
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-693
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Moderate Plaque Psoriasis; Severe Plaque Psoriasis; Plaque Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with Moderate to Severe Plaque Psoriasis: Subjects with Moderate to Severe Plaque Psoriasis in Greece

SUMMARY:
This study estimates the treatment goal achievement rate, depicts the implementation of the Progressive Psoriasis Initiative (PPI) recommendations regarding treatment modifications and transitioning, and assesses patient adherence and persistence with adalimumab therapy in the routine clinical practice in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis for at least 6 months, and moderate to severe disease course at the time of adalimumab treatment onset, defined as Body Surface Area (BSA) >10 or PASI >10 and DLQI >10
* Patients for whom the decision to prescribe therapy with adalimumab (Humira®) according to the locally approved summary of product characteristics (SmPC) has already been taken prior to their enrolment in the study and is clearly separated from the physician's decision to include the patient in the current study
* Patients with an available Psoriasis Area Severity Index (PASI) and Dermatology Life Quality Index (DLQI) scores at the start of adalimumab treatment
* Patients able and willing to provide written informed consent and to comply with the requirements of this study protocol
* Patients with a signed informed consent document

Exclusion Criteria:

* Patients should not have non-plaque forms of psoriasis (e.g., erythrodermic, guttate, or pustular)
* Patients for whom treatment with adalimumab has been initiated more than 2 weeks prior to their enrolment into the study
* Patients that meet any of the contraindications to the administration of the study drug according to the latest version of the locally approved SmPC
* Patients who have previously been exposed to adalimumab unless a period of at least 6 months from the last dose has elapsed
* Patients currently receiving treatment with any investigational drug/device/intervention or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with adalimumab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Moderate to Severe Plaque Psoriasis in Greece
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who will achieve the European Consensus Programme (ECP)-defined treatment goals at the end of the induction phase (i.e. 16 weeks post-treatment onset) | 16 weeks post-treatment
  Achievement of the treatment goals during the induction phase is defined as:
  * Treatment Success: i.e. >=75% Psoriasis Area Severity Index (PASI) score reduction OR
  * Intermediate Response with Dermatology Life Quality Index (DLQI) <=5: i.e. PASI score reduction >=50% but <75% with DLQI <=5.

SECONDARY OUTCOMES:
Proportion of participants achieving intermediate response | Up to 12 months
  Intermediate response is defined as participants with PASI score reduction >=50% but <75% compared to week 0 (baseline).
Proportion of participant achieving treatment success | Up to 12 months
  Treatment success rate is defined as participants with >=75% PASI score reduction compared to week 0 (baseline).
Proportion of participant with treatment failure | Up to 12 months
  Treatment failure is defined as participants with PASI score reduction <50% compared to week 0 (baseline).
Proportion of participants achieving the treatment goals | Up to 12 months
  According to the European Consensus Programme (ECP) guidelines, achievement of the treatment goals during the maintenance phase is defined as:
  * Treatment Success: i.e. >=75% Psoriasis Area Severity Index (PASI) score reduction compared to the time of therapy initiation (i.e. baseline) (or)
  * Intermediate Response with Dermatology Life Quality Index (DLQI) <=5: i.e. PASI score reduction >=50% but <75% compared to baseline, with DLQI <=5.
Time to the first missed dose during the study observation period | Up to 12 months
  Patient diary will be reviewed to assess this information

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (43):
- Greece (43):
  - General Univ Hosp "Attikon" /ID# 149517, Athens, Attica
  - Tzaneio general hospital of Piraeus /ID# 149518, Piraeus, Attica
  - General Uni hosp of Larissa /ID# 149688, Larissa, Thessaly
  - General Uni hosp of Larissa /ID# 151442, Larissa, Thessaly
  - PP of Konstantinos Tsaousis /ID# 149704, Amaliáda
  - PP of Maria Sifaki /ID# 149717, Arkalochóri
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 158934, Athens
  - PP of Michael Kakepis /ID# 149693, Athens
  - PP of Georgios Papadopoulos /ID# 149712, Athens
  - PP of Ioannis Krikellis /ID# 149715, Athens
  - PP of Markos Papakonstantis /ID# 149702, Athens
  - PP of Panagiotis Deligiannis /ID# 149708, Athens
  - Genl Hospital Andreas Syggros /ID# 149516, Athens
  - Genl Hospital Andreas Syggros /ID# 149687, Athens
  - PP of Ekaterini Galaterou /ID# 149713, Athens, AGIA Paraskeui
  - PP of Ioannis Papaggelopoulos /ID# 149703, Athens, Ampelokipi
  - PP of Antonios Seretis /ID# 149714, Athens, Chalandri
  - PP of Despoina Arnaoutoglou /ID# 149707, Athens, Glyfada
  - PP of Maria Loukatou /ID# 149706, Athens, Glyfada
  - PP of Eirini Stefanaki /ID# 149695, Athens, NEA Filadelfeia
  - PP of Pantelis Aronis /ID# 149705, Athens, NEA Smyrni
  - PP of Theognosia Vergou /ID# 149694, Athens, VARI
  - PP of Ioannis Mparkis /ID# 149711, Athens,neo Irakleio
  - PP of Vasilios Chatzakis /ID# 149718, Crete, Heraklion
  - PP of Kalliopi Karamanolaki /ID# 149720, Crete, Heraklion
  - PP of Vasiliki Tzirka /ID# 149722, Drama
  - Kontargiris, MD, Kalamata, GR /ID# 151444, Kalamata
  - Konstantopouleio General Hospi /ID# 149690, Nea Ionia
  - PP of Konstantinos Markakis /ID# 149723, Orestiáda
  - Rigatos, MD, Patra, GR /ID# 151446, Pátrai
  - University Gen Hosp of Patra /ID# 149691, Pátrai
  - PP of Chrysa Zisimou Politopou /ID# 149728, Stilís
  - PP of Aimilios Lallas /ID# 149721, Thessaloniki
  - PP of Pantelis Souvantzidis /ID# 149726, Thessaloniki
  - PP of Stelios Charalampidis /ID# 149727, Thessaloniki
  - PP of Georgios Chaidemenos /ID# 149724, Thessaloniki
  - General Hospital of Thessaloni /ID# 149692, Thessaloniki
  - Kallidis, MD, Thessaloniki, GR /ID# 151443, Thessaloniki
  - General Hospital of Thessaloniki George Papanikolaou /ID# 149515, Thessaloniki
  - Manousari, MD, Veroia, GR /ID# 151445, Véroia
  - PP of Prodromos Christoforidis /ID# 149730, Volos
  - General Hospital of Xanthi /ID# 149519, Xánthi
  - PP of Stathis Gkourvelos /ID# 149709, Xilokastro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-693.pdf